CLINICAL TRIAL: NCT00738205
Title: Evaluation of Convenience and Compliance of the Easypod™ Electronic Self-injector When Administering Saizen® Growth Hormone to Children With Growth Disorders
Brief Title: Evaluation of Convenience and Compliance of the Easypod™ Electronic Self-injector
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: Easypod
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Growth Hormone Deficiency; Turner Syndrome; Chronic Renal Failure; Small for Gestational Age
Keywords: Electronic device; Growth hormone treatment
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This is an international, multicenter study involving children treated with Saizen®, a growth hormone, who will be trained to use easypod, a new electronic injector and will complete a questionnaire after 12 week of use.

Both children naïve to growth hormone and dissatisfied with their current injection device will be recruited.

DETAILED DESCRIPTION:
An international, multicenter cross-sectional study (Observatoire des pratiques médicales®) involving a cohort of children treated with Saizen®, a growth hormone.

The study does not require any changes to the usual medical management of these patients and should not be considered detrimental to their physical or psychological integrity. No specific procedures or examinations will be requested, nor does the protocol require any particular treatment or follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Already treated patients who are dissatisfied with their current self-injection device, or naïve pediatric patients, in cases for which this indication is validated (growth hormone deficiency, Turner's syndrome, chronic renal failure, small-for-gestational age [SGA] patients, based on RCP)

Exclusion Criteria:

* Cases in which Saizen® is contra-indicated (based on local RCP)
* Children returning for consultation, who have not brought back their Easypod™ electronic self-injector.
* Children who are participating in a therapeutic trial, or who have done so in the 3-month period preceding their recruitment into this observational study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Overall, 834 children using the electronic auto-injector were recruited. Of these, 824 children were included in the evaluable population. Of the 824 evaluable children, 601 were treatment-naïve and 223 were treatment-experienced.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To assess children's compliance with the Saizen®, growth hormone treatment, following introduction of the new easypodTM self-injector, while comparing newly treated and previously treated children. | week 12

SECONDARY OUTCOMES:
To assess the acceptability of the new Easypod™ electronic injector for children following a growth hormone treatment regimen. | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Clément Olivier, MD, LMCC, Study Director — Merck Serono S.A., Geneva

REFERENCES:
- [Result] Bozzola M, Colle M, Halldin-Stenlid M, Larroque S, Zignani M; easypod survey study group. Treatment adherence with the easypod growth hormone electronic auto-injector and patient acceptance: survey results from 824 children and their parents. BMC Endocr Disord. 2011 Feb 4;11:4. doi: 10.1186/1472-6823-11-4. PMID 21294891